CLINICAL TRIAL: NCT06433505
Title: A Phase 1, Open-label, Two-Part Study to Evaluate the Pharmacokinetics, Metabolism and Excretion, and Absolute Bioavailability of BMS-986365 in Healthy Male Participants
Brief Title: A Study to Evaluate the Drug Levels, Metabolism and Excretion, and Absolute Bioavailability of BMS-986365 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA071-1005
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
Keywords: BMS-986365; Pharmacokinetics; Absolute Bioavailability; Healthy Male Volunteers; CC-94676; ADME

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental)
  Interventions: Drug: BMS-986365; Drug: [14C] BMS-986365
- Part B - Arm 1 (Experimental)
  Interventions: Drug: [14C] BMS-986409 + BMS-986410
- Part B - Arm 2 (Experimental)
  Interventions: Drug: [14C] BMS-986410 + BMS-986409

INTERVENTIONS:
Drug: BMS-986365 — Specified dose on specified days
  Arms: Part A
Drug: [14C] BMS-986365 — Specified dose on specified days.
  Arms: Part A
Drug: [14C] BMS-986409 + BMS-986410 — Specified dose on specified days
  Arms: Part B - Arm 1
Drug: [14C] BMS-986410 + BMS-986409 — Specified dose on specified days
  Arms: Part B - Arm 2

SUMMARY:
The objective of this study is to assess the pharmacokinetics (PK) and absolute bioavailability of BMS-986365 and to investigate the PK, metabolite profile, routes and extent of elimination, and mass balance of BMS-986365.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants as determined by no clinically significant deviations from normal in medical history, physical examination, 12-lead ECGs, or clinical laboratory determinations, as determined by the investigator
* Participants will require a left ventricular ejection fraction of > 50% at screening.
* Body mass index of 18.0 to 32.0 kg/m2, inclusive, at screening. Body mass index = weight(kg)/(height [m])2.

Exclusion Criteria:

* Any current or recent significant acute or chronic illness.
* Participants with a prior history of heart failure, ischemic heart diseases, serious cardiac arrythmias, or prolonged QTcF interval (> 450 ms) at screening.
* Current or recent (within 3 months of intervention administration) gastrointestinal disease that could affect the absorption of study drug including cholecystectomy. Mild gastroesophageal reflux (even if managed with avoidance of food triggers) is exclusionary.
* History of allergy to BMS-986365 or related compounds.

Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to Day 60
  Part A and B
Time of maximum observed concentration (Tmax) | Up to Day 60
  Part A and B
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to Day 60
  Part A and B
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC (INF)) | Up to Day 60
  Part A and B
Apparent terminal plasma half-life (T-HALF) | Up to Day 60
  Part A and B
Total body clearance (CLT) | Up to Day 15
  Part A
Apparent total body clearance (CLT/F) | Up to Day 60
  Part A and B
Mean residence time (MRT) | Up to Day 15
  Part A
Apparent volume of distribution (Vz) | Up to Day 15
  Part A
Apparent volume of distribution (Vz/F) | Up to Day 60
  Part A and B
Absolute bioavailability (F) | Up to Day 15
  Part A

SECONDARY OUTCOMES:
Number of participants with Adverse Events | Up to Day 60
  Part A and B
Number of participants with Serious Adverse Events | Up to Day 60
  Part A and B
Number of participants with AEs leading to discontinuation | Up to Day 60
  Part A and B
Number of participants with Vital sign abnormalities | Up to Day 60
  Part A and B
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 60
  Part A and B
Number of participants with physical examination abnormalities | Up to Day 60
  Part A and B
Number of participants with clinical laboratory abnormalities | Up to Day 60
  Part A and B

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Madison, Wisconsin, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com